CLINICAL TRIAL: NCT04515940
Title: Evaluation of the Acceptability (including Gastrointestinal Tolerance, Compliance and Palatability) of a High Energy Peptide Based Paediatric Oral Nutritional Supplement for Children Over 12 Months of Age
Brief Title: Acceptability and Tolerance Study of a High Energy Peptide Based Paediatric Oral Nutritional Supplement for Children
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: ONS peptide 1.5
Record Dates: First submitted 2020-03-06; First posted 2020-08-17 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Drug Tolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: acceptability, tolerance and palatability study — prospective acceptability study

SUMMARY:
This is an acceptability study (including gastrointestinal tolerance, compliance and palatability) of a high energy peptide based paediatric oral nutritional supplement for children over 12 months of age.

The acceptability data from a minimum of 15 participants will be collected in order to submit an application to the Advisory Committee on Borderline Substances (ACBS).

DETAILED DESCRIPTION:
Fifteen (15) participants, aged 12 months and over, requiring a high energy peptide based oral nutritional supplement drink for the dietary management.

The ACBS requirement for evaluable data on 15 participants has informed the trial's recruitment target; however, we may need to exceed this target if any patients give their consent to join the study but then decide not to participate in the study. Participants who join the study and begin using the product would count towards the recruitment total and their data would be included in a submission to the ACBS whether they complete the 7-day study period or not.

Each potential participant must meet all of the inclusion criteria and not meet any of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

I. Children aged 1 year and over who require 1-3 bottles of an oral nutritional peptide based supplement drink II. Children who require an oral nutritional supplement or who are already established on a nutritional supplement drink III. Children who require a nutritional supplement drink as bolus feeding via a feeding tube.

IV. Children being able to communicate views of acceptability V. Willingly given, written, informed consent from patient or parent/guardian. VI. Willingly given, written assent (if appropriate).

Exclusion Criteria:

I. Inability to comply with the study protocol, in the opinion of the investigator.

II. Contraindications to any feed ingredients (see nutritional table and ingredients list) III. Require a milk free diet IV. Children under the age of 12 months V. Emergencies

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: paediatric children 1- 10 years
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Day 7 from baseline
  Daily record via participant diary:
  1. Gastrointestinal tolerance:
     * Diarrhoea and / or constipation
     * Bloating and / or distension
     * Nausea and / or vomiting
     * Burping / flatulence / regurgitation
     * Abdominal discomfort / pain/ back arching/ crying
  2. Participant compliance:
     How many feeds taken and volume prescribed each day
  3. Acceptability
  Questionnaires to children and or parents for the evaluation of the acceptability and ease of use of the milk supplement drink Diarrhoea, constipation, bloating, distension, nausea, vomitting, burping, abdominal pain
Compliance | Day 7 from baseline
  volume suggested versus consumed

SECONDARY OUTCOMES:
weight in kg | Day 8 from baseline
  At baseline
height in meters | Day 8 from baseline
  At basline

CONTACTS AND LOCATIONS:
Overall Officials: Chris Smith, Principal Investigator — Nutrition and Dietetics
Locations (1):
- Nutrition and Dietetics, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No